CLINICAL TRIAL: NCT02572557
Title: A Prospective Evaluation of Spray Cryotherapy in Patients With Malignant and Benign Central Airway Disease
Brief Title: TruFreeze Cryotherapy Central Airway Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TruFreeze cryotherapy
Record Dates: First submitted 2015-10-02; First posted 2015-10-09 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Airway Obstruction
Keywords: Spray Cryotherapy
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spray cryotherapy using liquid nitrogen (Experimental): Device: TruFreeze Spray CryoTherapy Drug: Liquid nitrogen
  Interventions: Device: TruFreeze Spray CryoTherapy; Drug: Liquid nitrogen

INTERVENTIONS:
Device: TruFreeze Spray CryoTherapy — TruFreeze Spray CryoTherapy using liquid nitrogen
Drug: Liquid nitrogen — TruFreeze Spray CryoTherapy using liquid nitrogen

SUMMARY:
Rationale: Spray cryotherapy (SCT) using liquid nitrogen has been safely and effectively used in the esophagus, airways and pleura. Treatment with SCT for central airway stenosis may provide an effective, and more durable and perhaps safer alternative to the current therapeutic modalities.

Objectives:

1. To investigate the feasibility of using Spray cryotherapy (SCT) for the treatment of malignant and benign central airway disease.
2. To investigate the safety of using Spray cryotherapy (SCT) for the treatment of malignant and benign central airway disease.
3. To investigate the efficacy of using Spray cryotherapy (SCT) for the treatment of malignant and benign central airway disease.

Study design: This study will be a prospective, single arm, open label intervention study performed at the University Medical Center Groningen, The Netherlands Study population: The study population exists of 25 patients with malignant or benign central airway disease. Patients in which current treatment options are regarded to be suboptimal can be included in the study.

Intervention: TruFreeze Spray CryoTherapy

Main study parameter:

Feasibility is defined as being able to apply the SCT as planned in one, or more bronchoscopies according to the instructions for use (IFU).

Secondary study parameters:

Safety will be assessed by capturing all adverse events (AEs) that occur 1) during the SCT procedure, and 2) all AEs that occur until hospital discharge.

Efficacy will be measured using 1) patient reported outcomes (questionnaires), 2) percentage improvement in airway stenosis, 3) durability of treatment effect, 4) need to re-intervene with other therapies because of treatment failure.

Nature and extent of the burden, risks and benefit associated with participation.

Patients that will be recruited and participate in this prospective clinical trial have a severe central airway disease which is highly symptomatic for which current available therapies are either very difficult to perform, are hazardous, have no real benefit, or just simply not available yet. The current treatment risks of this patient group are high, especially in the patients where the airway patency is at risk. The main additional risk associated with the use of SCT is the occurrence of a pneumothorax. Patients participating will adhere to their current medical care, with the one addition of a voluntary follow-up bronchoscopy after SCT.

ELIGIBILITY:
Inclusion Criterium:

1. Presence of malignant or benign central airway disease where current treatment options are regarded to be suboptimal.

Exclusion Criteria:

1. Patient has an inability to tolerate bronchoscopy under general anaesthesia.
2. Compromised tissue (significant ulceration or mucosal break in the ablation area, any procedure or pre-existing condition has significantly reduced tissue strength or has significantly reduced the elasticity of the ablation area).
3. Airway diameter causing an anatomical flow resistance inhibiting N2 gas evacuation (Endotracheal tube or equivalent <8.5mm will be excluded).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of procedures in which SCT was applied as planned [Feasibility] | During bronchoscopy procedure
  Feasibility is defined as being able to apply the SCT as planned in one, or more bronchoscopies according to the instructions for use
Adverse events during procedure [Safety] | During bronchoscopy procedure
  Safety will be assessed by capturing all adverse events (AEs) that occur during the SCT procedure.
Adverse events during hospital admission [Safety] | Up to 5 days after treatment
  Safety will be assessed by capturing all adverse events (AEs) that occur until hospital discharge.

SECONDARY OUTCOMES:
Patient reported outcomes [Efficacy] | 4 weeks follow up
  Efficacy will be measured using patient reported outcomes (questionnaires).
Percentage improvement in airway stenosis [Efficacy] | 4 weeks follow up
  Efficacy will be measured by percentage improvement in airway stenosis.
Time in weeks of durability of initial improvement in airway stenosis[Efficacy] | 4 weeks follow up
  Efficacy will be measured by durability of treatment effect (time in weeks)
Number of patients with need to re-intervene [Efficacy] | 4 weeks follow up
  Efficacy will be measured by the need to re-intervene with other therapies because of treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen

REFERENCES:
- See also: Website of the bronchoscopic intervention center of the UMCG — http://www.bicumcg.nl